CLINICAL TRIAL: NCT03744936
Title: Decision Aids for Patients With Nonvalvular Chronic Atrial Fibrillation (DA4AFib)
Acronym: (DA4AFib)
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Victor Montori, MD, Prinicpal Investigator, Mayo Clinic
Other Study IDs: 18-007275
Record Dates: First submitted 2018-11-13; First posted 2018-11-19 (Actual); Results first posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-12

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nonvalvular Chronic Atrial Fibrillation (DA4AFib): Subjects who are scheduled for Nonvalvular Chronic Atrial Fibrillation (DA4AFib) treatment at Mayo Clinic Rochester and Mayo Clinic Health System sites in Minnesota
  Interventions: Other: Feedback

INTERVENTIONS:
Other: Feedback — Study team members will conduct interviews with subjects to gather feedback on Atrial Fibrillation experiences

SUMMARY:
The researchers are observing subject and clinician interaction in order to develop future education materials that will help patients and clinicians discuss atrial fibrillation and options to treat it.

ELIGIBILITY:
1. Must be 18 or older
2. Must have an appointment for Atrial Fibrillation
3. Must not have dementia
4. Must not have severe hearing or vision impairment Patients will be given a written consent Guests that accompany patients will be given an oral consent KER unit PAG members will be given an oral consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Encounters of subjects scheduled for AF (Atrial Fibrillation) treatment will be observed (by a study team member and/or using a video recording device) at Mayo Clinic Rochester and may be observed at Mayo Clinic Health System sites in Minnesota.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2020-02-06 (Actual); Study Completion 2020-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victor M Montori, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jones AE, McCarty MM, Cameron KA, Cavanaugh KL, Steinberg BA, Passman R, Kansal P, Guzman A, Chen E, Zhong L, Fagerlin A, Hargraves I, Montori VM, Brito JP, Noseworthy PA, Ozanne EM. Development of Complementary Encounter and Patient Decision Aids for Shared Decision Making about Stroke Prevention in Atrial Fibrillation. MDM Policy Pract. 2023 Jun 21;8(1):23814683231178033. doi: 10.1177/23814683231178033. eCollection 2023 Jan-Jun. PMID 38178866

RESULTS

PARTICIPANT FLOW:
Groups:
- Nonvalvular Chronic Atrial Fibrillation (DA4AFib): Subjects who were scheduled for Nonvalvular Chronic Atrial Fibrillation (DA4AFib) treatment at Mayo Clinic Rochester and Mayo Clinic Health System sites in Minnesota
  Study team members conducted interviews with subjects to gather feedback on Atrial Fibrillation experiences
Period: Overall Study
Arm/Group | Nonvalvular Chronic Atrial Fibrillation (DA4AFib)
Started | 34
Completed | 34 (34 patients)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Nonvalvular Chronic Atrial Fibrillation (DA4AFib)
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 13
Age, Continuous [Median (Full Range); unit: years] | 50 [21 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 33
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Interview Process
Description: The number of subjects to complete the interview process
Time Frame: baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Nonvalvular Chronic Atrial Fibrillation (DA4AFib)
Number analyzed (Participants) | 34
Participants | 34

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed.
Description: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed.
Arm/Group | Nonvalvular Chronic Atrial Fibrillation (DA4AFib)
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-01-24): https://cdn.clinicaltrials.gov/large-docs/36/NCT03744936/Prot_000.pdf
  • Informed Consent Form (2019-08-15): https://cdn.clinicaltrials.gov/large-docs/36/NCT03744936/ICF_001.pdf